CLINICAL TRIAL: NCT04396717
Title: A Phase 1, Sequential Cohort, Open-Label, Dose-Escalation Study of the Safety and CNS Exposure of Pritumumab in Patients with Brain Cancer
Brief Title: Safety Study of Pritumumab in Brain Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nascent Biotech (Industry)
Collaborators: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 08091967
Record Dates: First submitted 2020-04-29; First posted 2020-05-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Malignant Primary Brain Tumors; Brain Metastases, Adult
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Open label, non-randomized, 3+3 dose escalation to determine MTD, followed by exoansion to 6-12 patients to determine RP2D. Subjects will continue study treatment until progressive disease or unacceptable toxicity. Follow-up will occur until death or lost to follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pritumumab (Experimental): Dose Escalation phase (3+3 patients):
  Pritumumab administered sequentially as 1-hour IV infusion, on Day 1, 8, and 22 of each 28-day treatment cycle at: 1.6 mg/kg, 4.8 mg/kg, 8.0 mg/kg, 12.0 mg/kg, and 16.2 mg/kg, for a maximum of 6 cycles or progression or unacceptable toxicity.
  Expansion phase (6-12 patients): Pritumumab administered as 1-hour IV infusion, on Day 1, 8, and 22 of each 28-day treatment cycle at or below MTD for a maximum of 6 cycles or progression or unacceptable toxicity.
  Interventions: Biological: Pritumumab

INTERVENTIONS:
Biological: Pritumumab — Pritumumab IgG1 human monoclonal antibody

SUMMARY:
Pritumumab is a human IgG1 kappa antibody that binds to a malignant tumor associated antigen, ecto domain-vimentin (EDV) which is expressed in a variety of tumor cells. Pritumumab was shown to have relatively high reactivity with brain cancer cell lines, while no reactivity was demonstrated with normal neurons, astrocytes or fetal cerebral cells. Pritumumab has notable antibody-dependent cellular cytotoxicity (ADCC), brain tumor penetration and antitumor activity in nude mouse human xenograft models.

Primary Objectives

- To determine the safety and/or tolerability and the recommended Phase 2 dose (RP2D) of escalating, intravenously (IV) administered Pritumumab doses in patients with recurrent gliomas or with brain metastases.

Secondary Objectives

* To determine pharmacokinetics and pharmacodynamics of Pritumumab
* To identify preliminary signals of anti-tumor response to Pritumumab
* To explore disease-related, patient-reported outcomes

DETAILED DESCRIPTION:
This is an open-label, Phase 1, outpatient, dose escalation study of Pritumumab in patients with brain cancer who have failed prior therapy and have no other available options. In the first part of the study, escalating doses of Pritumumab of 1.6, 4.8, 8.0, 12.0, and 16.2 mg/kg will be administered in a sequential, safety-driven manner to eligible patients according to standard 3+3 scheme, as an 1-hour IV infusion on Days 1, 8, 15, and 22 of each 28-day treatment cycle. The dose levels may be modified upon obtained results. Once the maximum tolerated dose (MTD) is determined, an expansion cohort including 6-12 patients in selected tumor type at a dose equal or below to MTD is planned to determine the recommended Phase 2 dose (RP2D). A total of 42 patients may be administered with Pritumumab in this study.

Patients will be treated with Pritumumab for a maximum of 6 cycles or until cancer progression or unacceptable toxicity. Patients will be followed after treatment completion every four months or until death or lost to follow-up. Standard clinical, laboratory and functional assessments will be employed to monitor for safety, tolerability and tumor response, including blood sampling for clinical biochemistries, pharmacokinetics, CSF and tissue samples, at frequency specified by the protocol. Patient-reported outcomes will also be assessed.

ELIGIBILITY:
Inclusion Criteria Subjects must meet all of the inclusion criteria to participate in this study.

1. Ability to understand and the willingness to provide informed consent.
2. Diagnosis

   Histologically confirmed diagnosis of brain cancer:
   * glioblastoma (GBM),
   * anaplastic astrocytoma (AA),
   * anaplastic oligodendroglioma (AO),
   * anaplastic mixed oligoastrocytoma (AMO),
   * low grade gliomas,
   * brain metastases,
   * meningiomas, chordomas, medulloblastoma, craniopharyngiomas, pituitary tumors or
   * leptomeningeal metastases
3. Prior Therapy Has failed prior standard therapy including maximal safe surgical resection, radiation therapy (when appropriate for the specific cancer type), or systemic therapy or is intolerant of, or has refused other available therapies, but is still in need of therapy. No patients may receive Pritumumab prior to any surgery for their cerebral tumor
4. Progression/Recurrence Has progression of brain cancer and measurable disease by magnetic resonance imaging (MRI) or computed tomography (CT) scan.

   For leptomeningeal metastases, positive cytology is acceptable if imaging is not measurable.
5. Age Age ≥ 18 years.
6. Performance Status Karnofsky Performance Status ≥ 60% (see Appendix A). Subjects must have a life expectancy of equal to or greater than 8 weeks.
7. Organ and Marrow Function Requirements

   Hematology:
   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Hemoglobin ≥ 9.0 g/dL
   * White blood cell (WBC) count ≥ 3.0 x 109/L

   Biochemistry:
   * AST/SGOT and ALT/SGPT ≤ 5 x institution's ULN
   * Total bilirubin ≤ 3 x institution's ULN
   * Serum creatinine ≤ 2 x institution's ULN or 24-hour creatinine clearance ≥ 50 mL/min
   * Alkaline phosphatase (ALP) ≤ 3 x ULN unless considered tumor related
   * Estimated GFR > 50 mL/min

   Coagulation:
   * INR ≤ 1.4
   * PT/aPTT ≤ 1.2 x institution's ULN
8. Contraception All fertile females and any man with a partner of child-bearing potential agrees to use adequate contraception which will include two of the following: hormonal or barrier method of birth control, or abstinence prior to study entry, for the duration of study participation, and for 30 days following completion of therapy.
9. Although Pritumumab shows notable immunohistologic reactivity against active endometrial tissues, fertile female patients will be included in this study.

Exclusion Criteria Subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.

1. Current or anticipated use of other investigational agents.
2. Insufficient time for recovery from prior therapy:

   * less than 28 days from any prior cytotoxic investigational agent,
   * less than 14 days from any prior non-cytotoxic investigational agent,
   * less than 28 days from prior cytotoxic therapy (except 23 days from prior temozolomide at 5 day regimen and 14 days from prior temozolomide at daily regimen, 14 days from vincristine, 42 days from nitrosoureas, 21 days from procarbazine administration),
   * less than 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, targeted therapies (radiosensitizer does not count),
   * less than 7 days for immunotherapy agents, e.g., DCVax, Celldex, PD1, etc.
3. Less than 3 weeks from surgery or insufficient recovery from surgical-related trauma or wound healing.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pritumumab plus any patently atopic patients who have a history of having experienced an episode of allergic anaphylaxis.
5. Severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to receive study treatment (i.e., uncontrolled diabetes, chronic renal disease, chronic pulmonary disease or active, uncontrolled infection).
6. Known diagnosis of human immunodeficiency virus (HIV) infection.
7. Impaired cardiac function including any of the following:

   * Congenital long QT syndrome or a known family history of long QT syndrome;
   * History or presence of clinically significant ventricular or atrial tachyarrhythmias
   * Clinically significant resting bradycardia (< 50 beats per minute)
   * Inability to monitor the QT interval by ECG
   * QTc > 450 msec on baseline ECG. If QTc > 450 and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
   * Myocardial infarction within 1 year of starting study drug
   * Other clinically significant heart disease (e.g., unstable angina, congestive heart failure, or uncontrolled hypertension)
8. Any female patients who develop serious uterine hemorrhage during this study may need to be excluded from further treatment with Pritumumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 24 weeks
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE v.5.0 during first 24 weeks of treatment

SECONDARY OUTCOMES:
Intra-cranial Objective Response Rate | 2 months
  Intra-cranial objective response rate at 2 months as assessed by the Response Assessment in Neuro-oncology (RANO) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jose A. Carrillo, MD, Principal Investigator — One Hoag Drive Newport Beach, CA 92663, United States
Locations (2):
- United States (2):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Sharp Memorial Hospital, San Diego, California

IPD SHARING:
Plan to Share IPD: No